CLINICAL TRIAL: NCT05559970
Title: Effect of Inhalational Sedation on Mechanical Power in Mechanically Ventilated Patients: a Pilot Open-label Randomized Controlled Study
Brief Title: Inhalational Sedation and Mechanical Power
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 385/2565(IRB2)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation; Sedation; Mechanical Power; Lung Injury; ICU
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional sedation (Active Comparator): Conventional sedation receiving analgosedation with fentanyl
  Interventions: Drug: Convention sedation
- Inhalational sedation (Experimental): Inhalational sedation receiving isoflurane for sedation for 12 hours
  Interventions: Drug: Inhalational sedation

INTERVENTIONS:
Drug: Inhalational sedation — Inhalational sedation with isoflurane for 12 hours
  Arms: Inhalational sedation
Drug: Convention sedation — Conventional sedation receiving analgosedation with fentanyl
  Arms: Conventional sedation

SUMMARY:
Analgosedation is usually given to critically ill patients admitted in ICU. Fentanyl is the most common agent used for this purpose. For sedative agent, midazolam and propofol are commonly administered. However, too much sedation is apparently associated with increased duration of mechanical ventilation, prolonged ICU stay, and increased mortality.

In mechanically ventilated patients, mechanical power is the respiratory mechanic that can predict clinical outcomes including mortality in both ARDS and non-ARDS patients. Previous study demonstrated that sedating mechanically ventilated patients with propofol could decreased mechanical power. This was possibly associated with improved clinical outcomes in these patients.

At present, there is no clinical study investigating effects of inhalation sedation on mechanical power and clinical outcomes in mechanically ventilated patients.

DETAILED DESCRIPTION:
In the intensive care unit (ICU), sedation is used to improve comfort and tolerance during mechanical ventilation, invasive diagnostic and therapeutic interventions or nursing care. The most commonly used sedatives are intravenous benzodiazepines and propofol. These agents are associated with over-sedation in 40 to 60% of patients, which can lead to prolonged intubation, delirium and drug-induced hypotension. Volatile anesthetics are increasingly used for sedation in European and Canadian intensive care units that offer advantages of rapid drug on and off effects and clearance via pulmonary exhalation with no active metabolites. Delivery of volatile agents in the ICU can be simply performed using a small lightweight and portable anesthetic reflector so-called anesthesia conserving device. Compared with intravenous sedatives, volatile anesthetics may allow shorter time to extubation and can facilitate mental recovery.

In mechanically ventilated patients, a growing body of evidence suggests that the mechanical power (MP) plays an important role in the ventilator-induce lung injury (VILI) and prognosis in in both acute respiratory distress syndrome (ARDS) and non-ARDS patients. MP is the energy per unit time released to the respiratory system according to the tidal volume, PEEP, respiratory rate, and flow applied. In ARDS patients receiving invasive mechanical ventilation, high MP was associated an increased mortality. Moderate to deep sedation can inhibit the respiratory center and reduces the excessive respiratory drive, thereby reducing transpulmonary pressure and MP as well as probably reducing lung injury. The purpose of this study aims to investigate the effect of inhalation sedation on MP in mechanically ventilated patient admitted in the ICU. We hypothesize that MP in mechanically ventilated patients can be reduced by administering inhalational sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with age >18 years old; and
2. Patient who is admitted to the participating ICU; and
3. Patient who receives respiratory support with invasive mechanical ventilation via endotracheal tube < 12 hours prior to inclusion with anticipated duration of > 48 hours

Exclusion Criteria:

1. Patient with history or suspected history of malignant hyperthermia
2. Patient with evident or suspected increased intracranial pressure
3. Patient with high severity of illness whose ICU survival is not expected
4. Patient who refuses or patient whose proxy refuses to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in mechanical power | At 15 hours after intervention applied
  Change in mechanical power from Phase 1 to Phase 2 compared between 2 groups

SECONDARY OUTCOMES:
Change in oxygenation | At 15 hours after intervention applied
  Change in oxygenation from Phase 1 to Phase 2 compared between 2 groups
Change in respiratory mechanic | At 15 hours after intervention applied
  Change in respiratory mechanic from Phase 1 to Phase 2 compared between 2 groups
Change in serum interleukin 6 | At 15 hours after intervention applied
  Change in serum interleukin 6 from Phase 1 to Phase 2 compared between 2 groups
Change in serum C-reactive protein | At 15 hours after intervention applied
  Change in serum C-reactive protein from Phase 1 to Phase 2 compared between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Annop Piriyapatsom, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan of sharing individual participant data at this time.

REFERENCES:
- [Background] Grap MJ, Munro CL, Wetzel PA, Best AM, Ketchum JM, Hamilton VA, Arief NY, Pickler R, Sessler CN. Sedation in adults receiving mechanical ventilation: physiological and comfort outcomes. Am J Crit Care. 2012 May;21(3):e53-63; quiz e64. doi: 10.4037/ajcc2012301. PMID 22549581
- [Background] Jerath A, Parotto M, Wasowicz M, Ferguson ND. Volatile Anesthetics. Is a New Player Emerging in Critical Care Sedation? Am J Respir Crit Care Med. 2016 Jun 1;193(11):1202-12. doi: 10.1164/rccm.201512-2435CP. PMID 27002466
- [Background] Koutsogiannaki S, Shimaoka M, Yuki K. The Use of Volatile Anesthetics as Sedatives for Acute Respiratory Distress Syndrome. Transl Perioper Pain Med. 2019;6(2):27-38. doi: 10.31480/2330-4871/084. Epub 2019 Feb 21. PMID 30923729
- [Background] Bomberg H, Meiser F, Zimmer S, Bellgardt M, Volk T, Sessler DI, Groesdonk HV, Meiser A. Halving the volume of AnaConDa: initial clinical experience with a new small-volume anaesthetic reflector in critically ill patients-a quality improvement project. J Clin Monit Comput. 2018 Aug;32(4):639-646. doi: 10.1007/s10877-018-0146-z. Epub 2018 Apr 26. PMID 29700664
- [Background] Jerath A, Panckhurst J, Parotto M, Lightfoot N, Wasowicz M, Ferguson ND, Steel A, Beattie WS. Safety and Efficacy of Volatile Anesthetic Agents Compared With Standard Intravenous Midazolam/Propofol Sedation in Ventilated Critical Care Patients: A Meta-analysis and Systematic Review of Prospective Trials. Anesth Analg. 2017 Apr;124(4):1190-1199. doi: 10.1213/ANE.0000000000001634. PMID 27828800
- [Background] Landoni G, Pasin L, Cabrini L, Scandroglio AM, Baiardo Redaelli M, Votta CD, Bellandi M, Borghi G, Zangrillo A. Volatile Agents in Medical and Surgical Intensive Care Units: A Meta-Analysis of Randomized Clinical Trials. J Cardiothorac Vasc Anesth. 2016 Aug;30(4):1005-14. doi: 10.1053/j.jvca.2016.02.021. Epub 2016 Feb 23. PMID 27238433
- [Background] Coppola S, Caccioppola A, Froio S, Formenti P, De Giorgis V, Galanti V, Consonni D, Chiumello D. Effect of mechanical power on intensive care mortality in ARDS patients. Crit Care. 2020 May 24;24(1):246. doi: 10.1186/s13054-020-02963-x. PMID 32448389
- [Background] Costa ELV, Slutsky AS, Brochard LJ, Brower R, Serpa-Neto A, Cavalcanti AB, Mercat A, Meade M, Morais CCA, Goligher E, Carvalho CRR, Amato MBP. Ventilatory Variables and Mechanical Power in Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2021 Aug 1;204(3):303-311. doi: 10.1164/rccm.202009-3467OC. PMID 33784486
- [Background] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Background] Chiumello D, Gotti M, Guanziroli M, Formenti P, Umbrello M, Pasticci I, Mistraletti G, Busana M. Bedside calculation of mechanical power during volume- and pressure-controlled mechanical ventilation. Crit Care. 2020 Jul 11;24(1):417. doi: 10.1186/s13054-020-03116-w. PMID 32653011
- [Background] Spinelli E, Mauri T, Beitler JR, Pesenti A, Brodie D. Respiratory drive in the acute respiratory distress syndrome: pathophysiology, monitoring, and therapeutic interventions. Intensive Care Med. 2020 Apr;46(4):606-618. doi: 10.1007/s00134-020-05942-6. Epub 2020 Feb 3. PMID 32016537
- [Background] Jonkman AH, de Vries HJ, Heunks LMA. Physiology of the Respiratory Drive in ICU Patients: Implications for Diagnosis and Treatment. Crit Care. 2020 Mar 24;24(1):104. doi: 10.1186/s13054-020-2776-z. PMID 32204710
- [Background] Sahetya SK, Goligher EC, Brower RG. Fifty Years of Research in ARDS. Setting Positive End-Expiratory Pressure in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1429-1438. doi: 10.1164/rccm.201610-2035CI. PMID 28146639
- [Background] Xie Y, Cao L, Qian Y, Zheng H, Liu K, Li X. Effect of Deep Sedation on Mechanical Power in Moderate to Severe Acute Respiratory Distress Syndrome: A Prospective Self-Control Study. Biomed Res Int. 2020 Apr 11;2020:2729354. doi: 10.1155/2020/2729354. eCollection 2020. PMID 32351988